CLINICAL TRIAL: NCT04272372
Title: Multi Center Lymphedema Treatment Registry (LET) Study
Brief Title: Lymphedema Treatment Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Collaborators: Turkish Lymphedema Society (Unknown); The Breast Health Society, Turkey (Other)
Responsible Party: Principal Investigator, Sibel Eyigor, MD, Prof, Ege University
Other Study IDs: LET
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Lymphedema
Keywords: lymphedema; breast cancer; treatment
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Breast Neoplasms | interventions — Ketoprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Complete Decongestive Therapy
- Group 2: Complete Decongestive Therapy + PO Ketoprofen + Local ketoprofen gel
  Interventions: Drug: Ketoprofen
- Group 3: Complete Decongestive Therapy + Local Ketoprofen gel
  Interventions: Drug: Ketoprofen

INTERVENTIONS:
Drug: Ketoprofen — PO and local therapy
  Other Names: Ketoprofen topical
  Groups: Group 2; Group 3

SUMMARY:
Patients with breast cancer related lymphedema (clinical stage 0-2) will include in this study. Patients will take their demographic and clinical history and will evaluate with measurements of extremity volumes, body mass index, quality of life status and image studies (lymphoscintigraphy, Ultrasonography (USG), Indocyanine Green (ICG) Lymphograph or magnetic resonance imaging (MRI)) before and after the complete decongestive therapy. Outcome measurements such as limb volume, quality of life questionnaire and USG will repeat every 6,12,18, 24 months.

DETAILED DESCRIPTION:
Patients with breast cancer related lymphedema (clinical stage 0-2) will include in this study. Patients will take their demographic and clinical history and will evaluate with measurements of extremity volumes, body mass index, quality of life status and image studies (lymphoscintigraphy, USG, ICG or MRI) before and after the complete decongestive therapy (CDT). Outcome measurements such as limb volume, quality of life questionnaire and USG will repeat every 6,12,18, 24 months.

Group 1: CDT Group 2: CDT + PO ketoprofen +Local ketoprofen gel Group 3: CDT + Local ketoprofen gel

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Lymphedema more than 6 months
* Lymphedema stage 0-2
* Completed treatment (CT-RT)

Exclusion Criteria:

* Stage 3 lymphedema
* Cardiovasculary disease
* Hepatic disease
* Kidney disease
* Cerebrovascular event
* Metastasis
* Gastritis
* Infection
* Smoking
* Active cancer
* Bleeding history

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lyymphedema patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Limb Volume | 6,12,18, 24 months
  Volume measurements will take using ulnar styloid process as a index point, and circumferential measurements will take with 5 cm spaces from distal to the proximal. Using a computer programme (Limb Volumes Professional version 5.0), the total volume of the arm is calculate and record before and after the treatment for both arms.
  All patients' measurements before and after complete decongestive therapy will take by the same researcher. Volume changes will be evaluated at the 6th, 12th, 18th and 24.th months.

SECONDARY OUTCOMES:
Quality of Life status: Lymphedema Quality of Life Questionnaire-Arm (LYMQOL-ARM) | 6,12,18, 24 months
  LYMQOL-ARM questionnaire: The LYMQOL-Arm has been developed to assess the impact of lymphedema of the arms on the QoL of the patients. It consists of four domains with 28 items. These domains are symptoms, appearance, function, and mood. The answers were evaluated on a four-point Likert scale (1= not at all 2= a little, 3= quite a bit, 4= a lot). Each item received a score between 1 and 4, with higher scores indicating a worse QoL. Domain totals were calculated by adding the individual scores and dividing the total by the number of questions answered (If >50% of questions per domain were not answered this cannot be calculated
  *and =0). If the item was not scored and left blank or not applicable, this was scored with a 0. The four domains and their corresponding questions are: Function 1 (a-h), 2,3, Appearance 4,5,6,7,8 Symptoms 9,10,11,12,13,14 and Emotion 15,16,17,18,19,20. Overall QoL (Q21) is scored as the value marked by the patient, between 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Soran, Study Chair — University of Pittsburgh Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forte AJ, Boczar D, Huayllani MT, Lu X, McLaughlin SA. Pharmacotherapy Agents in Lymphedema Treatment: A Systematic Review. Cureus. 2019 Dec 5;11(12):e6300. doi: 10.7759/cureus.6300. PMID 31815082
- [Result] Rockson SG, Tian W, Jiang X, Kuznetsova T, Haddad F, Zampell J, Mehrara B, Sampson JP, Roche L, Kim J, Nicolls MR. Pilot studies demonstrate the potential benefits of antiinflammatory therapy in human lymphedema. JCI Insight. 2018 Oct 18;3(20):e123775. doi: 10.1172/jci.insight.123775. PMID 30333315
- [Result] Nakamura K, Radhakrishnan K, Wong YM, Rockson SG. Anti-inflammatory pharmacotherapy with ketoprofen ameliorates experimental lymphatic vascular insufficiency in mice. PLoS One. 2009 Dec 21;4(12):e8380. doi: 10.1371/journal.pone.0008380. PMID 20027220